CLINICAL TRIAL: NCT00804024
Title: Multi-center, Registry Trial of ClearWay™ RX Local Therapeutic Infusion Catheter for All Indications
Brief Title: ClearWay™ RX Registry Trial
Status: Completed | Type: Observational
Sponsor: Atrium Medical Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 20080711
Record Dates: First submitted 2008-12-05; First posted 2008-12-08 (Estimated); Last update posted 2013-04-19 (Estimated); Status verified 2013-04

CONDITIONS: Heart Diseases; Vascular Diseases
Keywords: Heart Diseases. Vascular Diseases.
MeSH Terms: conditions — Heart Diseases; Vascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day

GROUPS / COHORTS (1):
- ClearWay™ RX
  Interventions: Device: ClearWay™ RX Local Therapeutic Infusion Catheter

INTERVENTIONS:
Device: ClearWay™ RX Local Therapeutic Infusion Catheter — The ClearWay™ RX Local Therapeutic Infusion Catheter is a micro-porous PTFE balloon catheter designed for the localized infusion of various diagnostic and therapeutic agents into the coronary and peripheral vasculature.

SUMMARY:
The primary goal of this registry is to collect data regarding the use of the ClearWay RX Local Therapeutic Infusion Catheter for all indications.

DETAILED DESCRIPTION:
The registry will collect de-identified data regarding the indication for use, ease of use, drug perfusion, catheterization procedure details, success for intended use, and overall operator performance evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Subject required the use of the ClearWay Rx Local Therapeutic Infusion Catheter.

Exclusion Criteria:

* Subject not meeting the above inclusion criterion

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The ClearWay Rx Registry enrolled subjects who required the use of the ClearWay Rx Local Therapeutic Infusion Catheter.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2008-08; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
use, easy of use, drug perfusion, catheterization procedure details, success for intended use, and overall operator performance evaluation. | immediate

CONTACTS AND LOCATIONS:
Overall Officials: Ron Waksman, M.D., Principal Investigator — Medstar Health Research Institute
Locations (13):
- United States (13):
  - Escondido Cardiology Associates, Escondido, California
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Winter Haven Florida, Winter Haven, Florida
  - The Georgia Heart Center, Macon, Georgia
  - Clarian Health Partners Methodist Research Institute, Indianapolis, Indiana
  - Western Baptist Hospital, Paducah, Kentucky
  - Genesys Regional Medical Center, Grand Blanc, Michigan
  - Great Lakes Heart & Vascular Institute, Saint Joseph, Michigan
  - St.Mary's Duluth Clinic Health System, Duluth, Minnesota
  - Presbyterian Hospital Mid-Carolina Cardiology, Charlotte, North Carolina
  - Forsyth Medical Center-Cardiovascular Research, Winston-Salem, North Carolina
  - Good Samaritan Hospital, Lebanon, Pennsylvania
  - Virginia Cardiovascular Specialists, Richmond, Virginia